CLINICAL TRIAL: NCT04451577
Title: Epidemiologic, Clinical, Molecular Characteristics of Hospital Employees With or Without Covid-19 Infection: a Retrospective-prospective Cohort Study
Brief Title: Epidemiologic, Clinical, Molecular Characteristics of Hospital Employees With or Without Covid-19 Infection
Acronym: UNICODE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: UNICODE
Record Dates: First submitted 2020-06-25; First posted 2020-06-30 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: COVID

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — blood, pharyngeal swab, and for those hospitalized for COVID-19, also for the bronchoalveolar lavage and fecal samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- EMPLOYEES WITHOUT COVID-19 INFECTION: Humanitas group employees (including ICH, Humanitas University and Gavazzeni), and two validation cohorts.
  Negativity to COVOD-19 will be tested by peripheral blood samples every month for 6 months (or until seroconversion). If they are positive for anti- covid 19 antibodies, a test for positivity of the virus will be carried out. T
  Interventions: Other: No intervention
- EMPLOYEES WITH COVID-19 INFECTION: Humanitas group employees (including ICH, Humanitas University and Gavazzeni), and two validation cohorts.
  employees that are Sars-Cov-2 positive both symptomatic and asymptomatic, there will be at least 2 peripheral blood samples (5 and 3 ml) at every control visit until ascertained negativity. They will also undergo a pharyngeal swab for viral titers and microbiota analysis at enrollment and at negativity. In addition, a sample of saliva/sputum will be collected for most of the employees at positivity and at every control visit.
  For employees hospitalized but not requiring intensive care the following samples will be collected:
  * an aliquot of samples from the respiratory tract (e.g., bronchial aspirate, bronchoalveolar lavage) residual from the normal clinical practice
  * saliva/sputum
  * pharyngeal swab not used for diagnosis both at admission and at the first check up
  * blood sample in EDTA for plasma and peripheral blood mononuclear cell (PBMC)
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention, analysis of biological samples

SUMMARY:
The study cohort will be enrolled among all Humanitas group employees (including ICH, Humanitas University and Gavazzeni), and two validation cohorts. Participants will be asked consent for the research use of blood, pharyngeal swab, and for those hospitalized for COVID-19, also for the bronchoalveolar lavage and fecal samples. Biological samples will be used to perform cellular, microbial and molecular analyses aimed at better understanding the disease pathogenesis and the individual differences in susceptibility to the disease.

DETAILED DESCRIPTION:
The analysis will include:

* study the expression levels of molecules known to mediated viral infection, like the Angiotensin converting enzyme 2 (ACE2) and genetic variants in these genes, which could be related to susceptibility to the viral infection and/or to the severity of the clinical course of the disease
* compare the frequency of genetic variants potentially related with COVID-19 susceptibility/severity in different subgroups of patients, ranging from individuals positive for the virus but asymptomatic to individuals affected by COVID-19 with ARDS requiring admission to ICU
* germline DNA analysis to search for genetic factors predisposing or protecting against severe pulmonary affection in COVID-19 infected participants. To this aim DNA will be analyzed by a GWAS (Genome Wide Association Study) approach by using the GSA Illumina chip. The obtained data will also be used to try to develop a polygenic risk score to stratify individuals with a particularly high or low risk for severe disease course
* explore the contribution of rare variants by studying the exome
* sepsis and ARDS biomarkers developed at ICH (e.g. PTX3, sIL-1R2, MSF) analysis to address their prognostic potential in Covid-19 patients
* PBMC analysis by FACS to investigate the immunophenotype and correlate it to the clinical outcome
* microbiota analysis of residual BAL and pharyngeal swab to evaluate whether different microbial or metabolome profiles are associated to worsen disease or to protection
* plasma and saliva/sputum test for anti-SARS-Cov-2 antibodies (IgM, IgG, IgE and IgA) and for microbiota analysis

ELIGIBILITY:
Inclusion Criteria:

* 1. Individuals aged ≥ 18 years;

Exclusion Criteria:

* 1. Lack of informed consent according to local procedure per critically ill patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study cohort will be enrolled among all Humanitas group employees (including ICH, Humanitas University and Gavazzeni), and two validation cohorts
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Clinical response to COVID-19 | 36 months
  COVID-19 infection will be assessed by serological analysis of the presence of IgG anti-Covid-19 antibodies, an a subsequent pharyngeal swab. Symphtoms and possible hospitalization will be considered in clinical response.
Immunological response to COVID-19 | 36 months
  PBMC analysis by FACS to investigate the immunophenotype and correlate it to the clinical outcome (symptoms aggressiveness).
Genetic predisposition to COVID-19 | 36 months
  Genetic variants analysis potentially related with COVID-19 susceptibility/severity in different subgroups of patients, ranging from individuals positive for the virus but asymptomatic to individuals affected by COVID-19 with ARDS requiring admission to ICU
Microbiome-related response to COVID-19 | 36 months
  Microbiota analysis (using 16S rDNA sequencing technology) of residual BAL, pharyngeal swab, plasma and saliva/sputum to evaluate whether different microbial or metabolome profiles are associated to worsen disease or to protection

CONTACTS AND LOCATIONS:
Locations (1):
- Humanitas reseach hospital (ICH), Rozzano, Milan, Italy

IPD SHARING:
Plan to Share IPD: No